



| Use patient label Patient name: | CONSENT FORM |
|---------------------------------|--------------|
| DOB: | |
| Number: | |

## Immunity against RSV and influenza in a human experimental challenge model

| Principa | al investigator: Professor Peter Openshaw/Dr Christopher Chiu | Please initial |
|---|---|---|
| 1. | I confirm that I have read and understand the participant information sheet Version Twelve dated 12 <sup>th</sup> July 2018 for the above study and been given a copy to keep. I have had the opportunity to ask questions and have had these answered satisfactorily. | and tick |
| 2. | I understand that participation is voluntary, and that I am free to withdraw consent at any time, without giving any reason and without my medical care or legal rights being affected. | |
| 3. | I understand that sections of any of my medical notes and data collected during the study may be looked at by responsible individuals from Imperial College, Imperial College Healthcare NHS Trust or from regulatory authorities, where it is relevant to my taking part in this research. I give permission for these individuals to access my records. | |
| 4. | I understand that, after having my medical history taken, a physical examination and blood tests to make sure I am eligible, I will enter either the RSV or flu arm of the study. | |
| 5. | I agree to the use of my tissue samples in this research project, as described on the participant information sheet. I agree to my tissue samples being shared in some cases with collaborators (either UK or international) as long as they have local ethical approval. | |
| 6. | I agree to the use of my tissue samples in any future ethically-approved studies, including studies with UK or international collaborators | |
| 7. | I agree to my GP being informed of my participation in the study. | |
| 8. | I understand that if I enter the RSV or flu arm of the project I must remain in a residential facility at all times for a period of up to 10 nights during the study. | |
| 9. | I understand that if results of the study measurements of the immune response warrant further assessment of the correlation between the immune response and some genetic characteristics, these measurements will be performed. I agree to the use of my samples for these genetic measurements. | Yes No |

| Use patient label Patient name: | | | · |
|---------------------------------|------------------------|--------|---------|
| DOB: | | | |
| Number: | | | |
| 10. I agree to take part in | this research project. | | |
| Name of Participant | Signature | - Date | |
| Person taking consent | Signature | Date | Name of |

1 copy for participant; 1 copy for Principal Investigator; 1 copy to be kept with hospital notes.